CLINICAL TRIAL: NCT03411213
Title: Quantitative Assessment and Characterization of Microvascular Function Using Diffuse Optical Tomography Version
Brief Title: Quantitative Assessment and Characterization of Microvascular Function Using Diffuse Optical Tomography
Acronym: DOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STH18094
Record Dates: First submitted 2017-12-18; First posted 2018-01-26 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Atherosclerosis; Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vascular function (Experimental): Diffuse optical tomography detection of differences in vascular function between healthy volunteers and patients with proven heart disease or diabetes.
  Interventions: Device: diffuse optical tomography
- Coronary artery disease (Experimental): Diffuse optical tomography prediction of presence or severity of coronary artery disease on angiography.
  Interventions: Device: diffuse optical tomography

INTERVENTIONS:
Device: diffuse optical tomography — Optical tomography is a form of computed tomography that creates a digital volumetric model of an object by reconstructing images made from light transmitted and scattered through an object.

SUMMARY:
Atherosclerosis is accompanied by microvascular dysfunction (an impairment of blood vessels to dilate or constrict in response to demand). The ability to reliably measure microvascular dysfunction would help identify patients at risk of myocardial infarction and test new treatments. All existing measures of microvascular dysfunction suffer significant limitations.

Near Infrared Spectroscopy (NIRS) is an imaging method that uses an infrared light-source and detector (called optodes) to painlessly shines light into tissue and collect reflected light at different wavelengths. This data allows quantification of the amount of haemoglobin (blood) in the tissue and whether it is oxygenated or de-oxygenated.

Diffuse optical tomography (DOT) is a powerful analysis technique for data collected from multiple NIRH optodes. Unlike most NIRS studies that use a single pair of optodes and collects a single datapoint for each wavelength over time, DOT allows three-dimensional spatial reconstruction of haemodynamic and anatomic changes in a large region of tissue over time.

In preliminary work DOT had the potential to measure forearm reactive hyperaemia, a key indicator of microvascular function. Team will test whether DOT can detect differences between patients and healthy volunteers.

In this work, 30 patients will be recruited with type 2 diabetes, 30 patients who have had a previous myocardial infarction and 30 healthy volunteers. The Investigator will also recruit 50 patients who are on waiting lists for coronary angiography.

The DOT will be used to measure participants' microvascular function after brachial artery occlusion by a blood pressure cuff. The Investigator will then examine whether DOT can detect differences between healthy volunteers, diabetics, and patients with a previous heart attack, and whether DOT is able to predict existence of coronary artery disease on angiography. If successful, DOT can be developed for assessment of microvascular function to the point where it could be applied to clinical studies.

DETAILED DESCRIPTION:
Previous pilot studies have shown ability to collect promising data safely. In the following studies, the same study as in the pilot will be performed to apply the array of optodes to the surface of the arm. These emit light painlessly into the tissue and collect scattered light from the tissue. Inflation of a blood pressure cuff around the arm for 5 minutes, then deflate the cuff to allow blood flow back into the tissue. From the data gathered before, during and after the cuff is inflated, 3D reconstructions can be performed of HbO, HbR, and HbT changes in the forearm during and after arterial occlusion.

Study 1) Can DOT detect differences in vascular function between healthy volunteers and patients with proven heart disease or diabetes

This study will measure vascular function in patients with known heart disease (previous myocardial infarction) or diabetes and compare this to matched healthy volunteers. This will establish whether DOT can detect differences in vascular response between these groups. If so, then the method has the potential to be useful diagnostically or prognostically.

Potential participants will be approached by poster, or face to face in STH clinics and provided with the information sheet which participants will be asked to read at home. Participants will be given the opportunity to ask questions by email or telephone at any time afterwards. Participants will be asked to contact us if they are willing to participate.

Participants will be booked with an appointment to attend the Clinical Research Facility at Sheffield Teaching Hospitals (at least 24hrs after receiving the information sheet and having the chance to ask questions) for a visit of 30-45 minutes. Visits will be arranged in advance at a convenient time.

When participants attend, after agreeing to take part and signing a consent form, participants will take a seat in a private room. Participants will need to wear short sleeves, or roll their sleeves up. If necessary, the investigator can provide a gown to wear if the sleeves are too tight. The investigator will then do the following;

1. Record some details about medical history, height/weight, whether they take medications, date of birth, whether male or female.
2. Measure the blood pressure by briefly inflating a cuff around the upper arm.
3. Place an array of fibre optics on the surface of the forearm. Some jelly will be placed on the skin first, and the array will be held in place by a strap or tape. This is not painful.
4. After around 10 minutes of sitting quietly, the investigator will inflate a blood pressure cuff around the arm that the array is placed on. This will temporarily prevent blood entering or leaving the arm. This will feel tight and the arm may go numb. The investigator will keep the cuff inflated for five minutes, but the participant can ask for the cuff to be deflated at any time.
5. The investigator will then deflate the cuff, allowing blood back into the arm. After around 10 more minutes, the investigator will remove the cuff and array and the participant will be free to leave.

After the first assessment, the investigator will ask participants if they would be willing to attend for a second assessment where we would repeat the above measurements. This is to test how reproducible the measurements are in the same individual.

Study 2) Can DOT predict presence or severity of coronary artery disease on angiography?

This study will measure vascular function in patients awaiting diagnostic coronary angiography (either invasive or by CT), in whom it is not known whether or not coronary artery disease is present. Once the angiographic results are available the investigator will correlate vascular function measured by DOT with presence and severity of coronary artery disease to examine whether or not DOT identified

Potential participants will be approached by poster, or face to face in STH clinics and provided with the information sheet which participants will be asked to read. Participants will be given the opportunity to ask questions by email or telephone at any time afterwards. Participants will be asked to contact us if they are willing to participate.

Participants will be booked with an appointment to attend the Clinical Research Facility at Sheffield Teaching Hospitals (at least 24hrs after receiving the information sheet and having the chance to ask questions) for a visit of approximately 45 minutes. Visits will be arranged in advance at a convenient time.

When participants attend, after agreeing to take part and signing a consent form, particpants will take a seat in a private room. Participants will need to wear short sleeves, or roll their sleeves up. If necessary, the investigator can provide a gown to wear if the sleeves are too tight. the investigator will then do the following;

1. Record some details about medical history, whether they take medications, date of birth, whether male or female.
2. Measure the blood pressure by briefly inflating a cuff around the upper arm.
3. Place an array of fibre optics on the surface of the forearm. Some jelly will be placed on the skin first, and the array will be held in place by a strap or tape. This is not painful.
4. After around 10 minutes of sitting quietly, the investigator will inflate a blood pressure cuff around the arm that the array is placed on. This will temporarily prevent blood entering or leaving the arm. This will feel tight and the arm may go numb. The investigator will keep the cuff inflated for five minutes, but the participant can ask for the cuff to be deflated at any time.
5. The investigator will then deflate the cuff, allowing blood back into the arm. After around 10 more minutes, the investigator will remove the cuff and array and the participant will be free to leave.

Once the angiogram is performed (as part of their routine clinical care) the results will be reviewed by a clinically trained researcher. This will then be correlated with their vascular function measured by DOT to determine whether this can predict angiographic findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 of either sex
2. Ability to read and speak English to a level allowing understanding of the patient information and to give consent to participate
3. Diagnosed as type 2 diabetic for at least 12 months
4. No painful arms or health problems preventing blood pressure cuff inflation
5. No lymphoedema of the arm
6. Not diabetic or known to have suffered a myocardial infarction in the past

Exclusion Criteria:

Any patients that do not meet the above criteria will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Can diffuse optical tomography detect microvascular function? | 3 years from start date
  Measuring microvascular function with diffuse optical tomography

SECONDARY OUTCOMES:
Detecting differences in microvascular function in atherosclerosis | 3 years from start date
  Detecting differences in microvascular function using diffuse optical tomography between healthy people and those with atherosclerosis
Detecting differences in microvascular function in diabetes | 3 years from start date
  Detecting differences in microvascular function using diffuse optical tomography between healthy people and those with diabetes
Predicting coronary artery disease before angiography | 3 years from start date
  Predicting coronary artery disease before angiography using diffuse optical tomography

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Chico, Principal Investigator — University of Sheffield
Locations (1):
- Northern General Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marzilli M, Merz CN, Boden WE, Bonow RO, Capozza PG, Chilian WM, DeMaria AN, Guarini G, Huqi A, Morrone D, Patel MR, Weintraub WS. Obstructive coronary atherosclerosis and ischemic heart disease: an elusive link! J Am Coll Cardiol. 2012 Sep 11;60(11):951-6. doi: 10.1016/j.jacc.2012.02.082. PMID 22954239
- [Background] Tooke JE. Microvascular function in human diabetes. A physiological perspective. Diabetes. 1995 Jul;44(7):721-6. doi: 10.2337/diab.44.7.721. PMID 7789639
- [Background] Pyke KE, Tschakovsky ME. Peak vs. total reactive hyperemia: which determines the magnitude of flow-mediated dilation? J Appl Physiol (1985). 2007 Apr;102(4):1510-9. doi: 10.1152/japplphysiol.01024.2006. Epub 2006 Dec 14. PMID 17170205
- [Background] Charakida M, Masi S, Luscher TF, Kastelein JJ, Deanfield JE. Assessment of atherosclerosis: the role of flow-mediated dilatation. Eur Heart J. 2010 Dec;31(23):2854-61. doi: 10.1093/eurheartj/ehq340. Epub 2010 Sep 23. PMID 20864485
- [Background] Huang AL, Silver AE, Shvenke E, Schopfer DW, Jahangir E, Titas MA, Shpilman A, Menzoian JO, Watkins MT, Raffetto JD, Gibbons G, Woodson J, Shaw PM, Dhadly M, Eberhardt RT, Keaney JF Jr, Gokce N, Vita JA. Predictive value of reactive hyperemia for cardiovascular events in patients with peripheral arterial disease undergoing vascular surgery. Arterioscler Thromb Vasc Biol. 2007 Oct;27(10):2113-9. doi: 10.1161/ATVBAHA.107.147322. Epub 2007 Aug 23. PMID 17717291
- [Background] Mitchell GF, Parise H, Vita JA, Larson MG, Warner E, Keaney JF Jr, Keyes MJ, Levy D, Vasan RS, Benjamin EJ. Local shear stress and brachial artery flow-mediated dilation: the Framingham Heart Study. Hypertension. 2004 Aug;44(2):134-9. doi: 10.1161/01.HYP.0000137305.77635.68. Epub 2004 Jul 12. PMID 15249547
- [Background] Rubinshtein R, Kuvin JT, Soffler M, Lennon RJ, Lavi S, Nelson RE, Pumper GM, Lerman LO, Lerman A. Assessment of endothelial function by non-invasive peripheral arterial tonometry predicts late cardiovascular adverse events. Eur Heart J. 2010 May;31(9):1142-8. doi: 10.1093/eurheartj/ehq010. Epub 2010 Feb 24. PMID 20181680
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Dhawan AP, D'Alessandro B, Fu X. Optical imaging modalities for biomedical applications. IEEE Rev Biomed Eng. 2010;3:69-92. doi: 10.1109/RBME.2010.2081975. PMID 22275202
- [Background] Takagishi Y, Yamamura H. Purkinje cell abnormalities and synaptogenesis in genetically jaundiced rats (Gunn rats). Brain Res. 1989 Jul 17;492(1-2):116-28. doi: 10.1016/0006-8993(89)90894-9. PMID 2752293